CLINICAL TRIAL: NCT00556348
Title: Intravitreal Bevacizumab for Choridal Neovascularization Secondary to Age-Related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, MD, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JN-02-2007-ARVO
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Age Related Macular Degeneration
Keywords: bevacizumab; AMD; Complications; Visual acuity; OCt; Age Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — 1.25mg

SUMMARY:
To report the short term anatomic and visual acuity response after intravitreal injection of bevacizumab (Avastin, Roche, Rio de Janeiro, Brazil) in patients with choroidal neovascularization secondary to age-related macular degeneration.

DETAILED DESCRIPTION:
We conducted a retrospective study of 500 eyes with choroidal neovascularization secondary to age-related macular degeneration who were treated with at least two (initial and one month after) intravitreal injection of 1.25 mg bevacizumab and had a follow-up of at least 2 months. Patients underwent Snellen visual acuity testing, optical coherence tomography (OCT) imaging and ophthalmoscopic examination at baseline and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Age related macular degeneration with Juxtafoveal and Subfoveal CNVM: Recurrent CNVM following PDT and TTT with IVTA. Patient who could not afford PDT, Macugen or Lucentis which is FDA approved.
* Myopic CNVM, Idiopathic CNVM, Inflammatory CNVM and other conditions associated with CNVM.
* Refractory macular oedema due to vein occlusion, Pseudophakia, Clinically significant macular oedema (CSME) etc. that affects vision and does not respond adequately to usual treatment methods.
* Proliferative diabetic retinopathy, non-resolving vitreous haemorrhage with PDR.

Exclusion Criteria:

* Patients with poor compliance
* Patients with uncontrolled diabetes and hypertension or any other medical condition that increase the risk of complications like recent history of Stroke or myocardial infraction (< one year). (Physician clearance was obtained for all patients).
* Patients who had undergone major surgery 28 days before, were excluded from the study and it was also suspended prior to elective surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Vision change Anatomical changes (Regression of NVE, CNVM, reduction in macular thickness) Electrophysiological changes (ERG, VEP

SECONDARY OUTCOMES:
Ocular side effects (infection, RD, IOP rise, cataract)

CONTACTS AND LOCATIONS:
Overall Officials: Joao J Nassaralla, Jr, Principal Investigator — UnB and IOG